CLINICAL TRIAL: NCT00460824
Title: A Retrospective Review of Anti-HLA Antibodies and Donor Crossmatch Results as a Predictor of Pediatric Heart Transplant Outcomes
Brief Title: A Retrospective Review - Anti-HLA Antibodies
Status: Withdrawn | Type: Observational
Why Stopped: Not a Clinical trial. Retrospective Data review only.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Robert Bray, PhD, Professor, Emory University
Other Study IDs: IRB00003541
Record Dates: First submitted 2007-04-16; First posted 2007-04-17 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Congenital Disorders
Keywords: transplant; HLA antibodies matching; immunologic mismatching
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Transplant rejection following organ transplant occurs because the recipient's immune system attacks the transplanted organ. The recipients immune system recognizes the transplanted organ as foreign tissue and attempts to destroy it in the similar way that it attempts to destroy infectious agents such as bacteria and viruses. The human leukocyte antigen (HLA) system is a set of genes that is responsible for controlling an individuals' ability to tell the difference between an infectious agent and self tissue.

Differences in HLA genes between donors and recipients play a major part in influencing the rejection or acceptance of foreign tissue (i.e. transplanted organs). Due to time limitations in heart transplantation, HLA matching is not considered. It is unclear how individual HLA differences affect the recovery and expected lifespan of pediatric heart transplant recipients.

This study is designed to look at the donor-recipient matching and mismatching to determine if mismatching leads to more complications, shorter graft survival and, therefore, increased risk of death following pediatric heart transplantation.

DETAILED DESCRIPTION:
It is generally thought that immunologic mismatching in solid organ transplant will lead to increased rates of graft failure due to acute rejection in the short term and chronic rejection, or coronary vasculopathy in the longterm. Many studies in renal, pancreas and lung transplantation suggest favorable outcomes when HLA matching occurs and unfavorable outcomes when HLA mismatching occurs and circulating donor-specific antibodies are produced.

However, in heart transplantation this association is less clear. Advances in recognition and identification of HLA antibodies have resulted in more specific information regarding HLA mismatching and outcomes. This study is aimed at analyzing outcomes in pediatric heart transplant based on recipient-donor HLA incompatibility and the post-transplant production of donor-specific HLA antibodies.

Hypothesis:

1. HLA systems' genes class I & II matching results in a survival/rejection benefit in pediatric heart transplant recipients.
2. Mismatched transplants with donor-specific HLA antibodies have decreased overall survival.

A Multivariate Analysis of data will be performed by both Emory and Children's investigators and research support staff.

ELIGIBILITY:
Inclusion Criteria:

* heart transplants at Childrens Healthcare of Atlanta, Egleston Hospital
* transplants between July 1, 1988 through and including January 31, 2007
* complete HLA data
* survived more than 30 days after transplant

Exclusion Criteria:

* subjects undergoing retransplant

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: * heart transplants at Childrens Healthcare of Atlanta, Egleston Hospital
  * transplants between July 1, 1988 through and including January 31, 2007
  * complete HLA data
  * survived more than 30 days after transplant
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 1988-07

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bray, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States